CLINICAL TRIAL: NCT02773797
Title: Sedation and Physiologic Response to Intranasal Dexmedetomidine in Severe Chronic Obstructive Pulmonary Disease (COPD): A Randomized, Blinded, Placebo Controlled Crossover Trial
Brief Title: Placebo Controlled Evaluation of Sedation and Physiological Response to Intranasal Dexmedetomidine in Severe COPD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Dayton VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Nystrom02
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: COPD
Keywords: Sedation; Dexmedetomidine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IN-DEX 1.0 mcg/kg, intranasal saline (Placebo Comparator): Patients with clinically stable severe COPD will be randomized. Each group will participate in 3 drug study sessions separated by 7-14 days. Arm label "Intranasal-Dexmedetomidine (IN-DEX) intranasal 1.0 mcg/kg" will participate in 3 drug study sessions separated by 7-14 days. All drug study sessions will be conducted in a monitored acute care setting with medical staff in attendance. Sedation assessment and vital signs will be recorded at 15 minute and 5-15 minute intervals respectively, for a minimum of 3 hours.
  Interventions: Drug: IN-DEX 1.0 mcg/kg, intranasal saline
- IN-DEX, 1.5 mcg/kg intranasal saline (Placebo Comparator): Patients with clinically stable severe COPD will be randomized. Each group will participate in 3 drug study sessions separated by 7-14 days. Arm label "IN-DEX intranasal 1.5 mcg/kg" will participate in 3 drug study sessions separated by 7-14 days. All drug study sessions will be conducted in a monitored acute care setting with medical staff in attendance. Sedation assessment and vital signs will be recorded at 15 minute and 5-15 minute intervals respectively, for a minimum of 3 hours.
  Interventions: Drug: IN-DEX 1.5 mcg/kg, intranasal saline
- Placebo - Saline (Active Comparator): Patients with clinically stable severe COPD will be randomized. Each group will participate in 3 drug study sessions separated by 7-14 days. Arm label "Placebo - Saline" will participate in 3 drug study sessions separated by 7-14 days. All drug study sessions will be conducted in a monitored acute care setting with medical staff in attendance. Sedation assessment and vital signs will be recorded at 15 minute and 5-15 minute intervals respectively, for a minimum of 3 hours.
  Interventions: Drug: Placebo - Saline

INTERVENTIONS:
Drug: IN-DEX 1.0 mcg/kg, intranasal saline
  Other Names: precedex
  Arms: IN-DEX 1.0 mcg/kg, intranasal saline
Drug: IN-DEX 1.5 mcg/kg, intranasal saline
  Other Names: precedex
  Arms: IN-DEX, 1.5 mcg/kg intranasal saline
Drug: Placebo - Saline
  Arms: Placebo - Saline

SUMMARY:
A variety of medications have been used to treat the anxiety, discomfort, and fear associated with continuous and sudden episodic breathlessness in patients with advanced respiratory disease. Opioids and benzodiazepines, used alone or in combination, are commonly prescribed for this distressing symptom. Clinicians are concerned about the adverse effects of opioids, especially respiratory depression, so they frequently prescribe benzodiazepines. Recent studies have shown that benzodiazepine use is associated with adverse respiratory outcomes in older adults with Chronic Obstructive Pulmonary Disease (COPD). Dexmedetomidine may be an alternative to current drug therapies for breathlessness. Dexmedetomidine produces a dose dependent sedation, anxiolysis, and analgesia without respiratory depression or cognitive dysfunction.

The drug can be administered intranasally (IN-DEX) to induce light to moderate sedation of several hours duration.

The objective of the research is to assess the dose dependent safety and efficacy of intranasal dexmedetomidine compared to intranasal saline (placebo) in clinically stable patients with severe COPD. This will be accomplished in a staffed acute care setting with routine vital signs monitoring and continuous pulse oximetry. Patients will be assessed objectively and subjectively for their level of sedation by validated sedation scales.

The study is an extension of a similarly designed pilot study which did not include a placebo comparison. Results of the study will be helpful to design additional trials with intranasal dexmedetomidine in acutely symptomatic COPD patients, exertional dyspnea and exercise performance, and dyspnea treatment comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD (FEV1 < 50% predicted)
* Age 45-70
* American Society of Anesthesiologists (ASA) Class 3
* Body Mass Index < 35 kg/meter squared
* No prior history of adverse reactions to alpha 2 agonists (dexmedetomidine, clonidine)

Exclusion Criteria:

* known adverse reaction, allergy or hypersensitivity, to alpha 2 agonists
* Not nothing by mouth (NPO)
* ASA class >3
* Home oxygen therapy >2LPM by nasal cannula continuous use
* Any evidence of nasal mucosal inflammation, irritation, bleeding or ulceration
* Pregnancy, or possibility of pregnancy
* Coronary heart disease with stable or unstable angina
* Baseline heart rate <55 beats per minute
* Bradyarrhythmia, heart block, presence of pacemaker
* Congestive Heart Failure or known Cardiomyopathy (Ejection Fraction <40% by ECHO, MUGA, or myocardial perfusion imaging)
* Cor pulmonale
* Liver disease (hepatic transaminases > 2x upper limit of normal, cirrhosis, end stage liver disease)
* diagnosis of moderate to severe Obstructive Sleep Apnea
* currently enrolled in any other research study involving drugs or devices

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Modified Observer's Assessment of Alertness/Sedation Scale | every 15 minutes up to 5 hours after intranasal dexmedetomidine
Sedation Visual Analog Scale (VAS) | Every 15 minutes up to 5 hours after intranasal dexmedetomidine
Changes in Vital Signs | Every 5 minutes for 90 minutes, then every 15 minutes for up to 5 hours
  heart rate, noninvasive blood pressure, respiratory rate, continuous pulse oximetry

CONTACTS AND LOCATIONS:
Locations (1):
- Dayton VA Medical Center, Dayton, Ohio, United States